CLINICAL TRIAL: NCT06210516
Title: Effect of Respiratory Muscle Training on Diaphragm Function and Activity Performance in Subacute Ischemic Stroke Patients: A Single-blind Randomised-controlled Trial
Brief Title: Respiratory Muscle Training in Patients With Subacute Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sümeyye Akçay, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UniversityofHealthSciences
Record Dates: First submitted 2024-01-04; First posted 2024-01-18 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Subacute Stroke; Inspiratory Muscle Training
Keywords: Subacute Stroke; Ischemic; Respiratory Muscle Training; Ultrasonography; Activity Performance
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Intervention Model Description: A Randomised-controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Active Comparator): Inspiratory muscle training, aerobic training, breathing exercises neurophysiologic rehabilitation will be applied to the experimental group. This treatment program will be applied 5 sessions a week and totally 30 sessions (6 weeks).
  * Inspiratory muscle training
  * Aerobic training
  * Breathing Exercises
  * Neurophysiological Exercise Program
  Interventions: Device: PowerBreathe; Other: Conventional Physiotherapy
- Control Group (Active Comparator): The control group will receive aerobic training, breathing exercises and neurophysiological rehabilitation, excluding inspiratory muscle training.
  This treatment program will be applied 5 sessions a week and totally 30 sessions (6 weeks).
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Device: PowerBreathe — Primary Outcome Measurement:
  1. Maximal Inspiratory Pressure (MIP)
  Secondary Outcome Measurements:
  1. Chest circumference measurements
  2. Diaphragm movements and thickness (ultrasound)
  3. Hand grip strength (with a Jamar hand dynamometer)
  4. Motor Activity Log
  5. 6 Minute Walk Test (6MWT)
  6. Canadian Occupational Performance Measure
  7. Charlson Comorbidity Index
  Arms: Experimental Group
Other: Conventional Physiotherapy — Primary Outcome Measurement:
  1. Maximal Inspiratory Pressure (MIP)
  Secondary Outcome Measurements:
  1. Chest circumference measurements
  2. Diaphragm movements and thickness (ultrasound)
  3. Hand grip strength (with a Jamar hand dynamometer)
  4. Motor Activity Log
  5. 6 Minute Walk Test (6MWT)
  6. Canadian Occupational Performance Measure
  7. Charlson Comorbidity Index

SUMMARY:
Stroke, which can occur due to many different reasons and is one of the most common neurological conditions, is one of the leading causes of disability worldwide. The most common disorders that occur after stroke are motor disorders. In addition, these patients may be accompanied by respiratory problems such as changes in breathing patterns and decreased ventilation function. Respiratory problems are an important risk factor for the development of long-term mortality for both cardiovascular diseases and stroke. With all these changes, there is a serious decrease in the activity performance of the patients. While stroke rehabilitation focuses on motor function losses, problems in pulmonary functions do not receive the necessary attention. Evaluating and treating patients from every aspect in stroke rehabilitation will further increase the effectiveness of the treatments applied.

Ultrasonography (USG), which has been used in the field of healthcare for more than 40 years, works with a mechanism based on the principle of sound waves traveling and reflecting at different speeds in tissues of different densities. USG is a very useful and effective imaging method used by modern medicine as a part of examination and patient care, based on its advantages such as sound waves being harmless to living beings because they are non-ionizing, the image being real-time and being viewable at the time of the procedure, being a non-invasive method, and being inexpensive. This study will be included in the literature as an original study in terms of examining both the development of the patients and the effectiveness of the treatment in many aspects, with many parameters obtained by ultrasonography in subacute stroke patients who will receive respiratory muscle training.

DETAILED DESCRIPTION:
According to WHO, stroke, also known as cerebrovascular accident, is a neurological condition that results in rapidly developing loss of brain function as a result of a problem in the blood supply to the brain. Stroke, which ranks third among the causes of death, is one of the leading causes of disability. This neurological condition affects not only the periphery but also the respiratory muscles such as the diaphragm and intercostal muscles, causing respiratory weakness, changes in breathing patterns, and a decrease in respiratory volume. These changes in breathing lead to a decrease in physical activity and therefore limitation in daily living activities. The decrease in respiratory muscle strength results in an increase in morbidity and mortality due to decreased pulmonary function.

Pulmonary rehabilitation (PR) is the most common non-pharmacological treatment method for pulmonary diseases. PR has been studied extensively in patients with neuromuscular disease or spinal cord injury patients with restrictive pulmonary disease; However, studies in stroke patients with respiratory complications such as pneumonia are limited.

There are studies in the literature showing that respiratory muscle training applied after stroke has positive effects on various respiratory parameters.

In this study, the development of the pulmonary muscles with respiratory muscle training after stroke will be followed by ultrasound and functional tests, and the effect of this development on hand grip strength and activity performance, which is an indicator of general muscle strength, will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Having had a stroke for the first time,
* Being 18 years or older,
* Having an ischemic type stroke,
* At least 1 month has passed since the stroke,
* Modified Rankin Score ≥ 3,
* Ability to communicate,
* Agreeing to participate in the study.

Exclusion Criteria:

* Hemispatial neglect,
* Having a psychiatric disease,
* Having any breathing problems before the stroke,
* Not having any orthopedic, neurological or cardiopulmonary disease that would constitute a contraindication for the protocols to be applied,
* Being diagnosed with sarcopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure (MIP) | Change from pre-interventional MIP score at the end of the 30 sessions intervention that will be performed 5 days in a week at a total of 6 weeks.
  Maximal inspiratory pressure (MIP) is the most commonly used measure to evaluate inspiratory muscle strength. Measurement of MIP is a straightforward test in which individuals are asked to perform a forceful inspiration against an occluded mouthpiece. The advantages of this test are that it is noninvasive and performed quickly.

SECONDARY OUTCOMES:
Chest circumference measurements | Change from pre-interventional Chest circumference measurements at the end of the 30 sessions intervention that will be performed 5 days in a week at a total of 6 weeks.
  In order to evaluate chest mobility and breathing type, chest circumference measurements are taken from the axillary (4th rib level), epigastric (xiphoid process level) and subcostal (above the 11th and 12th ribs) regions using a tape measure.
Diaphragm movements and thickness (ultrasound) | Change from pre-interventional diaphragm movements and thickness (ultrasound) at the end of the 30 sessions intervention that will be performed 5 days in a week at a total of 6 weeks.
  Diaphragm ultrasonography is a non-invasive and portable imaging method that eliminates radiation exposure and does not require transfer of the person. Inspiratory thickness of the diaphragm (Ti), expiratory thickness of the diaphragm (Te), and mobility of the diaphragm will be measured.
Hand grip strength | Change from pre-interventional hand grip strength at the end of the 30 sessions intervention that will be performed 5 days in a week at a total of 6 weeks.
  Jamar hand dynamometer, which is accepted as the gold standard by the American Association of Hand Therapists (AETD) and has high validity and reliability in many studies, will be used to measure hand grip strength.
Motor Activity Log (MAL) | Change from pre-interventional MAL at the end of the 30 sessions intervention that will be performed 5 days in a week at a total of 6 weeks.
  Motor Activity Log is a measure used to assess the amount of use and quality of movement of paretic arms and hands in daily living activities for hemiparetic stroke patients. It consists of 30 items.
6 Minute Walk Test (6MWT) | Change from pre-interventional 6MWT at the end of the 30 sessions intervention that will be performed 5 days in a week at a total of 6 weeks.
  6 Minute Walk Test (6MWT) is a test adapted from the 12-minute Cooper test developed by Cooper and his colleagues in 1960 by the American Thoracic Society (ATS). 6MWT is defined as a submaximal test that can be easily applied to healthy or sick individuals and is considered as an indicator of exercise capacity and walking capacity as well as many cardiovascular diseases. 6MWT is referred to as the "Gold Standard" test of walking capacity.
Canadian Occupational Performance Measure (COPM) | Change from pre-interventional COPM at the end of the 30 sessions intervention that will be performed 5 days in a week at a total of 6 weeks.
  The Canadian Occupational Performance Measure (COPM) is a standard measurement tool used to determine an individual's activity performance problems and to measure the perception of performance change and performance satisfaction. In addition, COPM is an outcome measure that systematically helps identify activity performance problems that are important for the individual and rates improvements in these problems according to the individual's perspective. COPM consists of 3 parts: personal care (activities of daily living), productivity (education and work) and leisure (play, leisure activities, social participation).
Charlson Comorbidity Index | Change from pre-interventional Charlson Comorbidity Index score at the end of the 30 sessions intervention that will be performed 5 days in a week at a total of 6 weeks.
  Charlson comorbidity index was developed by Charlson et al. in 1987 to classify patients' comorbidities, determine their severity, and predict mortality rates. Each comorbidity of the patient is marked as "present" or "absent" and all scores are summed to obtain the total score. It is scored between 0-37.

CONTACTS AND LOCATIONS:
Overall Officials: Arsida Bajrami, M.D., Study Chair — IAU Medical Park Florya Hospital; Zuhal Kunduracılar, Prof. Dr., Study Chair — Saglik Bilimleri University; Dilber Karagözoğlu Coşkunsu, Ass.Prof., Study Chair — Fenerbahce University; Sümeyye Akçay, PT, Principal Investigator — Saglik Bilimleri University; Dudu Kübra Akyol, PT, Study Chair — IAU Medical Park Florya Hospital; Arzu Dinç Yavaş, M.D., Study Chair — IAU Medical Park Florya Hospital
Locations (1):
- Saglik Bilimleri University, Istanbul, Europe, Turkey (Türkiye)

REFERENCES:
- [Derived] Akcay S, Akyol DK, Erkut U, Karagozoglu Coskunsu D, Kunduracilar Z, Bajrami A, Dinc Yavas A. Effect Of Inspiratory Muscle Training on Diaphragm Function and Activity Performance in Subacute Ischemic Stroke Patients: A Single-Blind Randomized-Controlled Trial. Neurorehabil Neural Repair. 2026 Jan 27:15459683251412282. doi: 10.1177/15459683251412282. Online ahead of print. PMID 41589338